CLINICAL TRIAL: NCT00564343
Title: a Water Training Program to Improve Balance in Chronic Stroke Patients: Cross- Sectional Pre-Post Study Design
Brief Title: a Water Training Program to Improve Balance in Chronic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: itshak Melzer, Ben-gurion Univesity
Other Study IDs: sor425606ctil; ISRCTN4256
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Stroke Patients
Keywords: Balance; Water based training; Physical functioning; stepping behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ChSt, water training, Observation: Subjects suffer from chronic hemiplegia (a year or more post stroke) that upon questioning was judged to meet the following inclusion criteria: (a) able to stand independently 90 seconds; (b) able to walk 10 meters (with cane if necessary); (c) able to understand verbal instructions. The exclusion criteria will be: (a) Serious visual impairment; (b) Inability to ambulate independently (cane acceptable, walker not). (c) Severely impaired cognitive status (score less then 24 in Mini Mental State Examination). (d) Persons with impaired communication capabilities.
  Interventions: Other: water based training program to improve balance

INTERVENTIONS:
Other: water based training program to improve balance — The exercise group will meet on 24 occasions over a period of 12 weeks (2 times/week), 45 minute training session.

SUMMARY:
The proposed project is a case control study design. Subject's suffer from stroke willing to participate in the study will be shortly interviewed to assess eligibility according to the inclusion-exclusion criteria. Subjects suffer from chronic hemiplegia that upon questioning was judged to meet the following inclusion criteria: (a) able to stand independently 90 seconds; (b) able to walk 10 meters (with cane if necessary); (c) able to understand verbal instructions. The exclusion criteria will be: (a) Serious visual impairment; (b) Inability to ambulate independently (cane acceptable, walker not). (c) Severely impaired cognitive status (score less then 24 in Mini Mental State Examination). (d) Persons with impaired communication capabilities.

The whole project will be conducted over a period of 3 months. A total of 36 subjects will be assigned to water based exercise program. The exercise group will meet on 24 occasions over a period of 12 weeks (2 times/week). The subjects of the exercise group will be recruited from Sha'ar Ha'negev Swimming pool and from patients that get a Physical Therapy treatment Kupat Holim Clalit.

Gait and balance function will be tested in both groups with well established measuring techniques before and after the training period. The measuring techniques 1) Medical background variables. 2) Berg Balance Scale. 3) Late life Function and Disability Instrument. 4) Get up and go test - stand up and walk 3 meters turn around and walk back to the chair. 5) step execution test under single and dual task; 5) stability tests. 6) also fall will be monitored a year after the completion of the study. The water training intervention is performed on different levels where each level reflects different increasing demands on the postural control system. For example, the instructor can increase the difficulty of a certain water-exercise by instructing a participant to use less external support, close the eyes, decrease the support area (stand on one leg or narrow the stance, or on unstable surface). These "tools" allow the instructor to implement step exercises on a group level that are still challenging for each individual even if the skill level in the group varies. The water exercises also include perturbation exercises that trigger specific reflex-like balance responses. On each level the instructor can instantly modify an exercise to be more or less challenging for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects suffer from chronic hemiplegia (a year or more)
2. able to stand independently 90 seconds;
3. able to walk 10 meters (with cane if necessary);
4. able to understand verbal instructions.

Exclusion Criteria:

1. Serious visual impairment;
2. Inability to ambulate independently (cane acceptable, walker not).
3. Severely impaired cognitive status (score less then 24 in Mini Mental State Examination).
4. Persons with impaired communication capabilities.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The subjects of the exercise group will be recruited from Sha'ar Ha'negev Swimming pool and from patients that get a Physical Therapy treatment Kupat Holim Clalit.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

SECONDARY OUTCOMES:
Berg Balance Scale | fall will be monitored a year after the completion of the study.
Late life Function and Disability Instrument | fall will be monitored a year after the completion of the study
Get up and go test - stand up and walk 3 meters turn around and walk back to the chair | fall will be monitored a year after the completion of the study
Step execution test under single and dual task | fall will be monitored a year after the completion of the study
Stability tests | fall will be monitored a year after the completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dagan Shvartz, M.D., Principal Investigator — Ben-gurion University of the Negev, Beer-Sheva, Israel
Locations (1):
- SorokaUMC, Beersheba, Israel